CLINICAL TRIAL: NCT06880289
Title: PHASE II PROSPECTIVE RANDOMIZED TRIAL OF THE BOOST TREATMENT OF CHEMO-RADIOTHERAPY GUIDED BY PERFUSION MRI IMAGING ON HYPOXIC ZONES IN HEAD AND NECK CANCER
Brief Title: Chemo-Radiotherapy Boost Treatment Guided by Perfusion MRI on Hypoxic Zones in Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RS1308/20
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Tumors of the Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stIMRT standard IMRT regimen (Active Comparator): In this treatment arm, chemoradiotherapy will be administered at doses of 70 Gy, 63 Gy and 58.1 Gy will be administered to PTV1, PTV2 and PTV3 respectively in 35 fractions (5 fractions per week) with simultaneous integrated boost (SIB) technique.
  Chemotherapy will consist of i.v. cisplatin on days 1, 22, 43, at a dose of 100 mg/m2. Hydration and antiemetics are controlled according to the Institute guidelines.
  Interventions: Drug: Cisplatin IV on days 1, 22, 43, at a dose of 100 mg/m2
- deIMRT intensified IMRT regimen (Experimental): In the IMRT arm, the baseline HV dose (HV1) is further increased by 10% up to 77 Gy in 35 fractions (5 fractions per week) using SIB technique (2.2 Gy/fraction). Once the MR2 is performed at the 10th fraction, the hypoxic volumes (HV2) will be re-estimated and coregistered with the initial planning CT, if the HV2 is within the HV1, no change will be applied; if new hypoxic volumes are identified outside the initial HV1 volume, the plan will be adapted to boost these regions as well.
  Chemotherapy will consist of i.v. cisplatin on days 1, 22, 43, at a dose of 100 mg/m2. Hydration and antiemetics are controlled according to the Institute guidelines.
  Interventions: Drug: Cisplatin IV on days 1, 22, 43, at a dose of 100 mg/m2

INTERVENTIONS:
Drug: Cisplatin IV on days 1, 22, 43, at a dose of 100 mg/m2 — Chemoradiotherapy will be performed from day 1 to day 49 regardless of the arm.
  Other Names: Radioterapia 70 Gy, 63 Gy e 58.1 Gy

SUMMARY:
To assess and localize hypoxic tumor subregions both at baseline and during the second week of radiotherapy. And to hypothesize that an intensified IMRT regimen may ensure higher local response rates compared to the standard IMRT approach.

DETAILED DESCRIPTION:
A randomized, prospective, phase II study conducted with the aim of evaluating whether the strategy of overdosing hypoxic sub-regions of the primary tumor is associated with better local control compared to standard chemoradiotherapy for squamous cell carcinomas of the head and neck.

To evaluate whether side effects are influenced by the MRT approach. To search for initial (pre-treatment) hypoxic regions during treatment (at the 10th fraction of RT) in terms of volume and location. And finally to determine the prevalence and importance of pre-treatment hypoxic sub-regions and correlate the results with both clinical (primary site and tumor volume) and pathological (VEGF, EGFR and HIF-α expression in the primary tumor) characteristics.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed squamous cell carcinoma of the oropharynx, hypopharynx, or larynx;
* AJCC stage III or IV (cT2-4 N0-3 M0);
* specific informed consent.

Exclusion Criteria:

* Documented allergy to radiological contrast media or inability to receive contrast media due to concomitant pathology (e.g. renal);
* inability to receive radiotherapy (e.g. previous radiotherapy in the same region) and/or chemotherapy (inadequate bone marrow and/or liver and/or renal function);
* incomplete acquisition of MRI images;
* performance status 2 or more according to Zubrod;
* Previous invasive neoplasm (except skin cancer), except for neoplasms controlled for at least three years; non-invasive tumors (e.g. carcinoma in situ of the breast) are admitted even if diagnosed and treated in a period less than 3 years prior; patients with simultaneous or bilateral primary tumors are excluded;
* alcohol or drug abuse;
* legal incapacity or limited legal capacity;
* concomitant treatment with investigational drugs or participation in another clinical trial with use of investigational drugs within 30 days prior to screening for the study;
* documented hypersensitivity to study drugs or any of their excipients;
* pregnancy and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete response | 2 years
  Complete response is defined as complete disappearance (100%) of tumor at any site (primary and nodal) on both physical examination and imaging. Any site (primary or nodal) suspicious for residual disease on re-evaluation imaging or physical examination will be confirmed by pathology

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sanguineti, Doctor, Study Director — IRCCS National Cancer Institute
Locations (2):
- Italy (2):
  - IRCSS Regina Elena, Roma
  - "Regina Elena" National Cancer Institute, Rome